CLINICAL TRIAL: NCT03568071
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Repeated-dose Study to Evaluate the Efficacy, Safety, Tolerability,and PK/PD of Intravenously Administered MOR106 in Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Assess Efficacy, Safety, Tolerability and Pharmacokinetics (PK)/Pharmacodynamics (PD) of MOR106 in Subjects With Moderate to Severe Atopic Dermatitis
Acronym: IGUANA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: MOR106 clinical development in atopic dermatitis was stopped for futility
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOR106-CL-201; 2017-001142-10 (EudraCT Number)
Record Dates: First submitted 2018-05-31; First posted 2018-06-26 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort A - dose regimen A (Experimental): MOR106 will be administered as IV infusion. Subjects will receive repeated doses of MOR106 over a 12-week treatment period. A loading dose (dose regimen A) will be administered on Day 1.
  Interventions: Drug: MOR 106
- Cohort B - dose regimen B (Experimental): MOR106 will be administered as IV infusion. Subjects will receive repeated doses of MOR106 over a 12-week treatment period. A loading dose (dose regimen B) will be administered on Day 1.
  Interventions: Drug: MOR 106
- Cohort C - dose regimen C (Experimental): MOR106 will be administered as IV infusion. Subjects will receive repeated doses of MOR106 over a 12-week treatment period. A loading dose (dose regimen C) will be administered on Day 1.
  Interventions: Drug: MOR 106
- Cohort D - dose regimen D (Experimental): MOR106 will be administered as IV infusion. Subjects will receive alternating repeated doses of MOR106 or placebo over a 12-week treatment period. A loading dose (dose regimen D) will be administered on Day 1.
  Interventions: Drug: MOR 106
- Cohort E - dose regimen E (Experimental): MOR106 will be administered as IV infusion.Subjects will receive alternating repeated doses of MOR106 or placebo over a 12-week treatment period. A loading dose (dose regimen E) will be administered on Day 1.
  Interventions: Drug: MOR 106
- Placebo (Placebo Comparator): Subjects will receive repeated doses of placebo over a 12-week treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MOR 106 — The active pharmaceutical drug substance of MOR106 is a human immunoglobulin gamma-1 (IgG1) monoclonal antibody that binds with a high apparent affinity to human IL-17C.
  Arms: Cohort A - dose regimen A; Cohort B - dose regimen B; Cohort C - dose regimen C; Cohort D - dose regimen D; Cohort E - dose regimen E
Drug: Placebo — A sodium chloride infusion container with IV solution without addition of MOR106 drug product will be used as placebo in the proposed clinical study.
  Arms: Placebo

SUMMARY:
This is a Phase II, randomized, double-blind, placebo-controlled multicenter study of repeated doses of MOR106 administered as IV infusion. MOR106, is an antibody which is being developed as a treatment for diseases such as psoriasis and atopic dermatitis. An antibody is a protein that is made by the body in a defense reaction against viruses and bacteria or other small particles. In this case, MOR106 will act against IL-17C interleukin by binding to it. This way it could be possible to act against these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18-65 years of age (extremes included), on the day of signing informed consent form (ICF).
* Able and willing to give voluntary written informed consent and meet all of the inclusion criteria and none of the exclusion criteria before being enrolled in the study. The subjects must sign the informed consent form prior to any study-related procedures and agree to the schedule of assessments.
* A body mass index (BMI) between ≥18 and ≤30 kg/m².
* Diagnosis of chronic atopic dermatitis with at least 1 year since first diagnosis, as per the Hanifin and Rajka Criteria, fulfilling the following criteria:

  1. EASI ≥12 at screening and ≥16 at baseline (Day 1 pre-dose).
  2. Investigator's Global Assessment (IGA) score ≥3 (on the 0 to 4 IGA scale, in which 3 is moderate and 4 is severe) at screening and at baseline.
  3. Greater than or equal to 10% body surface area (BSA) of atopic dermatitis involvement at screening.
  4. Willingness to continue stable use of an additive free, basic, bland emollient twice daily for at least 7 days before baseline and throughout the study.
  5. Subject is a candidate for systemic therapy and has a history of inadequate response or has a contraindication to topical corticosteroids and/or topical calcineurin inhibitors before screening visit, as per investigator's opinion.
* Willing to adhere to the following contraceptive restrictions:

  1. Female subjects of childbearing potential must have a negative serum pregnancy test at screening, and a negative urine pregnancy test at baseline.
  2. Female subjects of childbearing potential must use a highly effective method of contraception from 28 days prior to the first dose of study drug, during the study, and for at least 24 weeks after the last dose of study drug.
  3. Non-vasectomized male subjects with a female partner of childbearing potential must agree to a highly effective form of contraception during the study, and for at least 24 weeks after last dose of study drug.
  4. All male subjects must agree to use a condom from the first dose of Investigational Medicinal Product (IMP), during the study and for at least 24 weeks after the last dose of IMP.

Exclusion Criteria:

* Known hypersensitivity to study drug ingredients or history of any significant allergic reaction to any drug as determined by the investigator, such as anaphylaxis requiring hospitalization.
* Prior treatment with MOR106.
* Positive serology for hepatitis B (positive hepatitis B surface [HBs] antigen and/or positive hepatitis core antibody [HBc]), or hepatitis C virus (HCV) antibody or any history of hepatitis from any cause with the exception of hepatitis A. Subjects who are immune to hepatitis B because of vaccination can be included.
* History of or current immunosuppressive condition (e.g., human immunodeficiency virus [HIV] infection), including history of invasive opportunistic infections (e.g., TB, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis), despite infection resolution or unusually frequent, recurrent, or prolonged infections, per investigator judgment.
* Subjects with a history of Varicella zoster virus who experienced any episode or recurrence of Herpes Zoster infection within 1 year of screening or ≥ one episode or Herpes Zoster within 1 year of screening must be excluded. (A history of Herpes simplex types 1 and 2 and vaginal candidiasis are permitted.)
* Pregnant or breast feeding female or subject is intending to become pregnant or breastfeed.
* Any concurrent illness, condition, disability, or clinically significant abnormality (including laboratory tests, ≥ New York Heart Association Classification (NYHA) III/IV) or clinically significant illness in the 3 months prior to initial study drug administration that, in the investigator's opinion, represents a safety risk for the subject's participation in the study, may affect the interpretation of clinical safety or efficacy data, or may prevent the subject from safely completing the assessments required by the protocol.
* Any of the following laboratory findings:

  1. White blood cell count <3.0 x 109 cells/L
  2. Neutrophil count <1.5 x 109 cells/L
  3. Platelet count <100 x 109 cells/L
  4. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 x upper limit of normal (ULN)
* History of malignancy within the past 5 years prior to screening with the exception of non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or of the breast, prostate cancer T1a or T1b using the TNM (tumour, nodes, metastasis) clinical staging system.
* Clinically significant abnormalities at the discretion of the investigator detected on vital signs or physical examination (other than atopic dermatitis) at screening or baseline (Day 1 pre-dose).
* History of eczema herpeticum in the last 12 months prior to screening.
* Subjects who have had an attenuated vaccination within 4 weeks of baseline or are expected to have one during the course of the study.
* Participation in another experimental therapy study within 5 times the half-life (if known) or 12 weeks (if not known) of the experimental therapy, prior to baseline, or current enrollment in any other interventional study.
* Having used any of the following treatments:

  1. Exposure to a biologic therapy for atopic dermatitis
  2. Immunosuppressive/ immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, interferon-gamma, azathioprine, methotrexate) within 4 weeks of baseline
  3. Phototherapy (ultraviolet [UV] B or psoralen and ultraviolet A [PUVA]) for atopic dermatitis within 4 weeks of baseline
  4. Treatment with topical corticosteroids or topical calcineurin inhibitors within 2 weeks of baseline
  5. Treatment with biologics (for non atopic dermatitis indications within 5 half-lives (if known) or 12 weeks prior to baseline (if unknown)
  6. Regular use (more than 2 visits per week) of a tanning booth/parlour within 4 weeks of screening
* Active chronic or acute infection requiring treatment with systemic (oral, SC or IV) antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals, within 4 weeks of baseline, or clinical signs of infective eczema within 1 week before baseline. Note: subjects may be rescreened after infection resolves.
* Investigator, research assistant, pharmacist, study coordinator, or other staff or relative thereof, who is directly involved in the conduct of the study.
* Not able to manage the electronic diary (e-diary) as per assessment of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Percent change in Eczema Area and Severity Index (EASI) score. | From baseline to Day 85
  To assess the clinical efficacy of repeated IV doses of MOR106 as assessed by percentage change from baseline in EASI score at Day 85 visit. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Proportion of subjects who achieve ≥50% overall improvement in Eczema Area and Severity Index (EASI) score. | From baseline to Day 85
  To assess the clinical efficacy of repeated IV doses of MOR106. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve ≥50% overall improvement in Eczema Area and Severity Index (EASI) score. | At Day 1
  To assess the clinical efficacy of repeated IV doses of MOR106. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve ≥50% overall improvement in Eczema Area and Severity Index (EASI) score. | At Day 15
  To assess the clinical efficacy of repeated IV doses of MOR106. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve ≥50% overall improvement in Eczema Area and Severity Index (EASI) score. | At Day 29
  To assess the clinical efficacy of repeated IV doses of MOR106. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve ≥50% overall improvement in Eczema Area and Severity Index (EASI) score. | At Day 43
  To assess the clinical efficacy of repeated IV doses of MOR106. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve ≥50% overall improvement in Eczema Area and Severity Index (EASI) score. | At Day 57
  To assess the clinical efficacy of repeated IV doses of MOR106. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve ≥50% overall improvement in Eczema Area and Severity Index (EASI) score. | At Day 71
  To assess the clinical efficacy of repeated IV doses of MOR106. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve an Investigators' Global Assessment (IGA) score of 0 or 1. | At Day 85
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve an Investigators' Global Assessment (IGA) score of 0 or 1. | At Day 1
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve an Investigators' Global Assessment (IGA) score of 0 or 1. | At Day 15
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve an Investigators' Global Assessment (IGA) score of 0 or 1. | At Day 29
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve an Investigators' Global Assessment (IGA) score of 0 or 1. | At Day 43
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve an Investigators' Global Assessment (IGA) score of 0 or 1. | At Day 57
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve an Investigators' Global Assessment (IGA) score of 0 or 1. | At Day 71
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve Investigators' Global Assessment (IGA) score reduction of ≥2. | At Day 85
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve Investigators' Global Assessment (IGA) score reduction of ≥2. | At Day 1
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve Investigators' Global Assessment (IGA) score reduction of ≥2. | At Day 15
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve Investigators' Global Assessment (IGA) score reduction of ≥2. | At Day 29
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve Investigators' Global Assessment (IGA) score reduction of ≥2. | At Day 43
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve Investigators' Global Assessment (IGA) score reduction of ≥2. | At Day 57
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Proportion of subjects who achieve Investigators' Global Assessment (IGA) score reduction of ≥2. | At Day 71
  To assess the clinical efficacy of repeated IV doses of MOR106.The IGA is an assessment scale to determine severity of atopic dermatitis and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Percent change in Scoring Atopic Dermatitis (SCORAD) score. | From baseline to Day 85
  To assess the clinical efficacy of repeated IV doses of MOR106. The SCORAD evaluates the extent of atopic dermatitis and ranges between 0 and 103. Higher values represent a worse outcome.
Percent change in Scoring Atopic Dermatitis (SCORAD) score. | At Day 1
  To assess the clinical efficacy of repeated IV doses of MOR106. The SCORAD evaluates the extent of atopic dermatitis and ranges between 0 and 103. Higher values represent a worse outcome.
Percent change in Scoring Atopic Dermatitis (SCORAD) score. | At Day 15
  To assess the clinical efficacy of repeated IV doses of MOR106. The SCORAD evaluates the extent of atopic dermatitis and ranges between 0 and 103. Higher values represent a worse outcome.
Percent change in Scoring Atopic Dermatitis (SCORAD) score. | At Day 29
  To assess the clinical efficacy of repeated IV doses of MOR106. The SCORAD evaluates the extent of atopic dermatitis and ranges between 0 and 103. Higher values represent a worse outcome.
Percent change in Scoring Atopic Dermatitis (SCORAD) score. | At Day 43
  To assess the clinical efficacy of repeated IV doses of MOR106. The SCORAD evaluates the extent of atopic dermatitis and ranges between 0 and 103. Higher values represent a worse outcome.
Percent change in Scoring Atopic Dermatitis (SCORAD) score. | At Day 57
  To assess the clinical efficacy of repeated IV doses of MOR106. The SCORAD evaluates the extent of atopic dermatitis and ranges between 0 and 103. Higher values represent a worse outcome.
Percent change in Scoring Atopic Dermatitis (SCORAD) score. | At Day 71
  To assess the clinical efficacy of repeated IV doses of MOR106. The SCORAD evaluates the extent of atopic dermatitis and ranges between 0 and 103. Higher values represent a worse outcome.
The number of incidents of Treatment-Emergent Adverse Events (TEAEs), Adverse Event of Special Interest (AESIs), Serious Adverse Events (SAEs), and discontinuations due to Adverse Events (AEs). | From screening up to Day 197/early discontinuation (ED) visit
  To assess the safety and tolerability of repeated IV doses of MOR106.
Characterization of the MOR106 immunogenetic profile. | From baseline through Day 197/ED visit
  To assess the immunogenicity of repeated IV doses of MOR106.
MOR106 (AUC0-inf) | From baseline through Day 197/ED visit
  To characterize the PK of repeated IV doses of MOR106.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Timmis, MBChB MICR, Study Director — Galapagos NV
Locations (53):
- Germany (16):
  - Fachklinik Bad Bentheim, Department of Dermatology, Bad Bentheim
  - Korsearch. Studienzentrum, Berlin
  - Charite, Universitätsmedizin Berlin, Centrum 12, Klinik für Dermatologie, Venerologie und Allergologie, Berlin
  - Hautarztpraxis im Jahrhunderthaus, Bochum
  - Hauttumorzentrum Ruhr- Universität Bochum, Bochum
  - RuhrDerm - Studienzentrum der Gemeinschaftspraxis für Dermatologie, Venerologie, Allergologie, Phlebologie, Bochum
  - Elbe Klinikum Buxtehude, Buxtehude
  - Universitätsklinikum Frankfurt, Klinik für Dermatologie, Frankfurt
  - SCIderm GmbH (a company of TFS group), Hamburg
  - Universitätsklinikum Heidelberg, Hautklinik, Heidelberg
  - Institut für Entzündungsmedizin, Lübeck
  - Clinical research center (CRC), Department of Dermatology, Mainz
  - Technical University Munich, Department of Dermatology, Munich
  - Klinik und Poliklinik der Dermatologie und Allergologie der Universität München, München
  - University Hospital of Muenster, Dpt. of Dermatology, Münster
  - Haut- und Lasercentrum Potsdam, Potsdam
- Hungary (5):
  - Budai Irgalmasrendi Kórház (St. John Hospital), Budapest
  - Semmelweis Egyetem Bőrgyógyászati Klinika, Budapest
  - Bács-Kiskun Megyei Kórház Bőrgyógyászati Osztály, Kecskemét
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház, Miskolc
  - Szegedi Egyetem Bőrgyógyászati és Allergológiai Klinika, Szeged
- Poland (27):
  - CERMED, Bialystok
  - Antoni Jurasz Universiti Hospital Nº1, Bydgoszcz
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - A-DERM-SERWIS NZOZ , Przychodnia Specjalistyczna, Częstochowa
  - Centrum Badań Klinicznych PI-House, Gdansk
  - Gyncentrum, Katowice
  - Centrum Medyczne ALL-MED, Krakow
  - Diamond Clinic, Krakow
  - Medical Center Dietla 19, Krakow
  - NZOZ Centrum Medyczne proMimed, Krakow
  - ETG Łódź, Lodz
  - Prywatny Gabinet Lekarski Urszula Chyrchel-Paszkiewicz, Lublin
  - Samodzielny Publiczny Szpital Kliniczny nr 1 Katedra i Klinika Dermatologii, Wenerologii i Dermatologii Dziecięcej, Lublin
  - Labderm sc Beata Bergler-Czop Barbara Sido-Bergler, Ossy
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Ostrowieckie Centrum Medyczne, Ostrowiec Świętokrzyski
  - KLIMED Marek Klimkiewicz, Piotrkow Trybunalski
  - Centrum Badan Klinicznych S.C., Poznan
  - Centrum Medyczne Grunwald, Poznan
  - Clinical Research Center Sp. z o.o. Medic-R Spółka Komandytowa, Poznan
  - ETG Skierniewice, Skierniewice
  - Centrum Medyczne AMED, Warsaw
  - Clinical Research Group, Warsaw
  - ETG Warszawa, Warsaw
  - 4HEALTH, Wroclaw
  - Dobrostan, Wroclaw
  - KLIMED Marek Klimkiewicz, Łomża
- University Hospital Bratislava, Bratislava, Slovakia
- United Kingdom (4):
  - Whipps Cross Hospital, Leytonstone
  - Plymouth Hospitals NHS Trust, Plymouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Royal Hallamshire Hospital, Sheffield
  - The Royal London Hospital, Whitechapel